CLINICAL TRIAL: NCT04656444
Title: Parental Compliance After Telephone Triage Advice During and After Confinement During the COVID-19 Epidemic in France
Acronym: COVIDTEL
Status: Withdrawn | Type: Observational
Why Stopped: obsolete study
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Other Study IDs: 20-HPNCL-03
Record Dates: First submitted 2020-12-04; First posted 2020-12-07 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- phone call to emergency department

SUMMARY:
Novel Coronavirus disease 2019 (COVID-19) outbreak seriously challenges worldwide health care systems. The current climate of anxiety due to COVID-19 and home confinement limiting access to emergency departments (ED) have induced an increase of phone calls to the emergency call center "15" medical advices.

To determine if a pediatric telephone triage protocol may improve patient's pathways during COVID-19 outbreak, parental compliance is assessed after telephone advice, during and after home confinement (the end of home confinement in France was on May 11th 2020).

From 14th April 2020 to 7th June 2020, all calls received by the platform of telephone calls at Children's Lenval Hospital during open hours and open days are collected. For each call, symptoms are recorded by trained physicians and trained residents using a telephonic triage tool through a directed interview. A medical orientation is recommended to parents at the end of their call. Follow-up are conducted 2 to 4 days after with their consent by telephone interview in order to evaluate their compliance

DETAILED DESCRIPTION:
Novel Coronavirus disease 2019 (COVID-19) outbreak seriously challenges worldwide health care systems. The current climate of anxiety due to COVID-19 and home confinement limiting access to emergency departments (ED) have induced an increase of phone calls to the emergency call center "15" for medical advices.

So far, Lenval Hospital pediatric ED didn't have a standardized telephonic triage protocol fitted to COVID-19 epidemic. Therefore, a telephonic triage tool is created as a decision support system in order to help physicians in regulating patient's pathways and in providing standardized medical advices.

To determine whether a pediatric telephone triage protocol may improve patient's orientation during COVID outbreak, parental compliance is assessed after telephone advice, during and after home confinement (the date of end of home confinement in France is 11th May 2020).

From 14th April 2020 to 7th June 2020, all calls received by the platform of telephone calls at Children's Lenval Hospital during open hours and open days are collected. For each call, symptoms are recorded by trained physicians and trained residents of the pediatric emergency department (PED) using a telephonic triage tool through a directed interview. A medical orientation is recommended to parents at the end of their call. Follow-up are conducted 2 to 4 days after with their consent by telephone interview in order to evaluate their compliance. Whatever the medical orientation given to parents, the investigators were able to visit PED in case of worsening of their child's condition or whenever they would feel the need a physical examination

Questioning parents about clinical condition of their child without a clinical look is challenging: on the one hand, clinical status of any sick child may change quickly; In the other hand, parents may not be reliable in evaluating their child's condition according to their level of concern. COVID-19 outbreak context may exacerbate parental anxiety and therefore induce inappropriate behavior.

Parents was considered as "non compliant" if they haven't followed the orientation initially given by the physician after telephone triage. They was considered as "compliant" (1) if they have respected the recommended orientation or (2) if they have had to bring their child at pediatric emergencies because of a worsening of his condition in the next 48 hours of the first call. In this specific case, to determine if the consultation at pediatric ED was necessary, the investigators recorded all resources utilization used and final orientation decided after visiting the ED. Thus, worsening of a child condition was defined as prescription of any diagnostic act and/or on-site therapeutic and/or hospitalization.

This study would allow to evaluate the applicability and the utility of a formalized telephone triage protocol fitted to COVID-19 epidemic, performed by trained medical staff in a Children's Hospital. Consequently, the investigators would be able to extend its use after the COVID outbreak period

ELIGIBILITY:
Inclusion Criteria:

Calls received by the platform of telephone calls at Children's Lenval Hospital on working days during working hours: Monday to Friday, 08h30-18h30, and Saturday 08h30-12h30

Exclusion Criteria:

Calls received during the weekends or holidays. Calls received outside working hours.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients calling the emergency department during working hours and days: Monday to Friday from 8:30 a.m. to 6:30 p.m. and Saturday morning between 8:30 a.m. and 12:30 p.m.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
parental compliance | at 24 hours post inclusion
  Compliance will be assessed by comparing the path defined by the doctor during the phone call and the orientation actually decided by the parents within 24 hours of the first phone call.

SECONDARY OUTCOMES:
parental anxiety | at 24 hours post inclusion
  The impact of advice given during a phone call on parental anxiety is assessed by comparing the level of anxiety between the first and second call (scale of 1, (not worried) to 5 (worried) )

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Pédiatrique de Nice CHU Lenval, Nice, France